CLINICAL TRIAL: NCT01263717
Title: Effects of Growth Hormone Releasing Hormone on Fat Redistribution, Cardiovascular Indices, and Growth Hormone Secretion in HIV Lipodystrophy
Brief Title: Effects of Growth Hormone Releasing Hormone in HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007p-000638
Record Dates: First submitted 2010-12-16; First posted 2010-12-21 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: HIV; HIV Lipodystrophy
Keywords: HIV; lipodystrophy; tesamorelin; Egrifta; growth hormone releasing hormone
MeSH Terms: conditions — Lipodystrophy | interventions — tesamorelin; Growth Hormone-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tesamorelin (Experimental): Tesamorelin (growth hormone releasing hormone) 2mg daily given subcutaneously x 6 months during randomized phase, followed by 6 months of open-label tesamorelin at same dose
  Interventions: Drug: tesamorelin
- Placebo (inactive injection) (Placebo Comparator): Placebo 2mg daily given subcutaneously for the first 6 months of the study, followed by 6 months of tesamorelin (growth hormone releasing hormone) 2mg daily during an open label phase
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tesamorelin — Tesamorelin (growth hormone releasing hormone) 2mg daily given by subcutaneous injection x 6 months during randomized phase, followed by 6 months of open-label tesamorelin at same dose
  Other Names: Egrifta, growth hormone releasing hormone, TH9507
  Arms: Tesamorelin
Drug: placebo — Placebo 2mg daily given by subcutaneous injection for the first 6 months of the study, followed by an open-label phase of 6 months of tesamorelin (growth hormone releasing hormone) treatment, 2mg daily given by subcutaneous injection
  Arms: Placebo (inactive injection)

SUMMARY:
HIV-infection and its treatment are often associated with an increase in belly fat, as well as abnormal cholesterol and problems metabolizing sugar. People with HIV infection and increased belly fat often have decreased growth hormone (GH) levels. Low GH levels may contribute independently to increased belly fat and to increased cardiovascular risk through effects on sugar metabolism, inflammation, and other mechanisms. Tesamorelin, a growth hormone releasing hormone (GHRH) analogue, has been shown to to reduce belly fat in patients with HIV-associated abdominal fat accumulation. However, the effects of tesamorelin on fat accumulation in the liver and muscle, sugar metabolism, and cardiovascular health are not yet known. The current study is designed to determine the effects of tesamorelin treatment on fat accumulation in the muscle and liver, insulin sensitivity and sugar metabolism, and markers of cardiovascular health including blood vessel thickness (carotid intima media thickness [cIMT]) and markers of inflammation in the body. The investigators hypothesize that tesamorelin will decrease fat accumulation in the liver and muscle and will decrease markers of inflammation, with either neutral or beneficial effects on glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65
2. Previously diagnosed HIV infection
3. Stable antiviral regimen for at least 12 weeks prior to enrollment
4. WC>95 cm and WHR>0.94 for male, WC>94 cm and WHR>0.88 for female occurring in the context of treatment for HIV disease
5. Subjective evidence of at least one of the following recent changes, occurring during the treatment of HIV disease: increased abdominal girth, relative loss of fat in the extremities, or relative loss of fat in the face
6. For female subjects 40yo or older, negative mammogram within one year of baseline

Exclusion Criteria:

1. Use of anti-diabetic agents, Megace, testosterone or any steroid use within 6 months of the study. Stable use of testosterone (> 6 mos) at dose equivalent to 200 mg IM q 2 weeks or < 10g/day to skin will be permitted.
2. Use of GH or GHRH within the past 6 months
3. Change in lipid lowering or antihypertensive regimen within 3 months of screening
4. Fasting blood sugar > 126 mg/dL, SGOT > 2.5 times ULN, HgB < 12.0 g/dL, creatinine > 1.4 mg/dL, CD4 count < 200
5. Severe chronic illness or active malignancy or history of pituitary malignancy or history of colon cancer
6. For men, history of prostate cancer or evidence of prostate malignancy by PSA > 5 ng/mL
7. Prior history of hypopituitarism, head irradiation or any other condition known to affect the GH axis
8. For women, positive urine hCG
9. Oral contraceptives, depo provera or combined progesterone-estrogen injections, transdermal contraceptive patches, estrogen or progestin coated IUD's within 6 months of the study.
10. Routine MRI exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clip.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Stanley TL, Feldpausch MN, Oh J, Branch KL, Lee H, Torriani M, Grinspoon SK. Effect of tesamorelin on visceral fat and liver fat in HIV-infected patients with abdominal fat accumulation: a randomized clinical trial. JAMA. 2014 Jul 23-30;312(4):380-9. doi: 10.1001/jama.2014.8334. PMID 25038357
- [Derived] Braun LR, Feldpausch MN, Czerwonka N, Torriani M, Grinspoon SK, Stanley TL. Fibroblast growth factor 21 decreases after liver fat reduction via growth hormone augmentation. Growth Horm IGF Res. 2017 Dec;37:1-6. doi: 10.1016/j.ghir.2017.10.002. Epub 2017 Oct 7. PMID 29031905

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Started | 28 | 26
Baseline Visit | 28 | 22
Completed | 23 | 20
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tesamorelin | Placebo (Inactive Injection) | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [46 to 54] | 53 [49 to 58] | 51.5 [46 to 56.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 24 | 18 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 14 | 34
  Black | 6 | 3 | 9
  Hispanic | 1 | 3 | 4
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: Liver Fat
Description: Hepatic fat as measured by magnetic resonance (MR) spectroscopy, and expressed by normalizing lipid to water and expressing as a percent (lipid-to-water percent).
Time Frame: 6 months
Population: All available data were used; data were not available for some subjects. Data from 1 patient who was discontinued between the 3 and 6mo visits for adverse event are included. These data were obtained at a termination visit.
Measure: Median (Inter-Quartile Range); unit: Change in hepatic lipid-to-water %
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 19
Change in hepatic lipid-to-water % | -2.0 [-6.4 to 0.1] | 0.9 [-0.6 to 3.7]

2. Primary Outcome: Visceral Adipose Tissue
Description: Change in visceral adipose tissue area as measured by single-slice computed tomography (CT) scan at the L4 vertebra.
Time Frame: 6 months
Population: Data from 1 patient who was discontinued between the 3 and 6mo visits for adverse event are included. These data were obtained at a termination visit.
Measure: Mean (95% Confidence Interval); unit: change in cm^2 after 6 months
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 24 | 20
change in cm^2 after 6 months | -34 [-53 to -15] | 8 [-14 to 30]

3. Secondary Outcome: Intramyocellular Lipid
Description: Intramyocellular lipid (IMCL) as measured by magnetic resonance (MR) spectroscopy of the calf. Soleus IMCL normalized to creatinine (IMCL/Cr based on areas determined by spectroscopy) was measured. The change over 6 months is reported.
Time Frame: 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Change in ratio of IMCL/Cr
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 23 | 20
Change in ratio of IMCL/Cr | -1.7 [-3.9 to 0.7] | -0.2 [-5.2 to 5.5]

4. Secondary Outcome: Endogenous Growth Hormone Secretion
Description: Endogenous growth hormone (GH) concentrations measured by overnight frequent blood sampling every 20 minutes. Mean overnight GH concentration is given.
Time Frame: 6 months
Population: All available data were used; data were not available for some subjects.
Measure: Median (Inter-Quartile Range); unit: Change in ng/mL
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 21 | 15
Change in ng/mL | 0.35 [0.15 to 0.57] | -0.01 [-0.07 to 0.06]

5. Secondary Outcome: Insulin Sensitivity
Description: In a subgroup of 1/2 of the subjects, euglycemic hyperinsulinemic clamp will be performed to assess insulin-stimulated glucose uptake. Insulin stimulated glucose uptake (M) calculated using the method of DeFronzo is shown.
Time Frame: 6 months
Population: All available data were used; data were not available for some subjects.
Measure: Mean (95% Confidence Interval); unit: Change in mg/kg/min
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 10 | 9
Change in mg/kg/min | 0.4 [-1.2 to 1.9] | 0.7 [-0.6 to 2.1]

6. Secondary Outcome: HbA1c
Description: Hemoglobin A1c.
Time Frame: 6 months
Population: All available data were used; data were not available for one subject.
Measure: Mean (95% Confidence Interval); unit: Change in %
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 20
Change in % | 0.20 [0.04 to 0.36] | 0.02 [-0.07 to 0.1]

7. Secondary Outcome: Insulin Like Growth Factor 1 (IGF-I)
Description: Insulin Like Growth Factor 1 (IGF-I).
Time Frame: 6 months
Population: All available data were used; data were not available for one subject.
Measure: Mean (Standard Deviation); unit: Change in ng/mL
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 20
Change in ng/mL | 79 (92) | 7 (62)

8. Secondary Outcome: Lipid Panel
Description: Fasting lipids. Triglyceride value is given.
Time Frame: 6 months
Population: All available data were used; data were not available for one subject.
Measure: Median (Inter-Quartile Range); unit: Change in triglyceride, mg/dL
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 20
Change in triglyceride, mg/dL | -25 [-68 to 8] | -10 [-33 to 8]

9. Secondary Outcome: Carotid Intimal Medial Thickness (cIMT)
Description: Carotid Intimal Medial Thickness (cIMT).
Time Frame: 6 months
Population: All available data were used.
Measure: Mean (95% Confidence Interval); unit: Change in mm
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 23 | 20
Change in mm | -0.03 [-0.07 to -0.00] | -0.00 [-0.03 to 0.03]

10. Secondary Outcome: Glucose Tolerance
Description: Glucose tolerance as measured by standard oral glucose tolerance test. 2-hour glucose is given.
Time Frame: 6 months
Population: All available data were used; data were not available for some subjects.
Measure: Mean (95% Confidence Interval); unit: Change in 2-hour glucose, mg/dL
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 18
Change in 2-hour glucose, mg/dL | -1 [-18 to 15] | -8 [-24 to 8]

11. Secondary Outcome: Adiponectin
Description: adiponectin.
Time Frame: 6 months
Population: All available data were used. Data were not available for 1 subject.
Measure: Median (Inter-Quartile Range); unit: Change in ng/mL
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 22 | 20
Change in ng/mL | 0 [-515 to 1159] | 0 [-1030 to 515]

12. Secondary Outcome: Hemostatic Markers
Description: Tissue plasminogen activator (tPA) and plasminogen activator inhibitor-1 (PAI-1) measured in serum.
Time Frame: 6 months
Population: Please note that we do not have data for these markers (neither PAI1 or tPA) because we did not have adequate funds to assess these.
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 month randomized portion of study
Arm/Group | Tesamorelin | Placebo (Inactive Injection)
Serious Adverse Events (participants affected / at risk) | 3/28 | 3/22
Other Adverse Events (participants affected / at risk) | 25/28 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tesamorelin (N=28) | Placebo (Inactive Injection) (N=22)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0) — exacerbation of existing congestive heart failure
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — pneumonia requiring hospitalization
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — diagnoses of basal cell carcinoma in 2 patients, both of whom had history of basal cell carcinoma in past
esophageal myotomy (Gastrointestinal disorders) | 0 (0) | 1 (1) — Planned Heller myotomy requiring post-procedure hospitalization
cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1) — acute cerebrovascular accident
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tesamorelin (N=28) | Placebo (Inactive Injection) (N=22)
injection site bruising (Skin and subcutaneous tissue disorders) | 10 | 11
paresthesia (Nervous system disorders) | 6 | 1
erythema at injection site (Skin and subcutaneous tissue disorders) | 4 | 2
joint pain (Musculoskeletal and connective tissue disorders) | 4 | 4 — arthralgia
stinging of skin (Skin and subcutaneous tissue disorders) | 3 | 0 — stinging at injection site
muscle pain (Musculoskeletal and connective tissue disorders) | 3 | 0 — myalgia
hyperglycemia (Endocrine disorders) | 2 | 2
edema (Blood and lymphatic system disorders) | 2 | 1
sinusitis (Infections and infestations) | 2 | 1

LIMITATIONS AND CAVEATS:
Please note that we intended to collect and analyze data on PAI1 and tPA but we did not have sufficient funds to do this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No